CLINICAL TRIAL: NCT05263804
Title: CoHort of Patients to Identify Biological and Imaging markerS of CardiovascUlar Outcomes in Stroke
Brief Title: CoHort of Patients to Identify Biological and Imaging markerS of CardiovascUlar Outcomes in Stroke - HIBISCUS-STROKE II
Acronym: HIBI STROKE II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL20_1003
Record Dates: First submitted 2021-01-18; First posted 2022-03-03 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-01

CONDITIONS: Ischemic Stroke
Keywords: Ischemic stroke; Stroke; Bio-collection; Imaging markers; Biomarkers; Clinical outcomes; Myocardial damages
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort group (Other): Patient over 18 with an ischemic stroke
  Interventions: Other: Collection of blood samples and MRI imaging in order to create a bio- and imaging-collection
- Ancillary study group (Experimental): Patient over 18 with an ischemic stroke
  Interventions: Other: Cardiac MRI with gadolinium injection - Ancillary Study

INTERVENTIONS:
Other: Collection of blood samples and MRI imaging in order to create a bio- and imaging-collection — No intervention. Collection of blood samples and MRI imaging in order to create a bio- and imaging-collection
  Arms: Cohort group
Other: Cardiac MRI with gadolinium injection - Ancillary Study — Collection of blood samples and MRI imaging in order to create a bio- and imaging-collection. 100 patients are expected in this group, for each of them, specific cardiac MRI with gadolinium injection will be done at day 6. Moreover, those 100 patients will follow the same visit schedule as the patients in the cohort group.
  Arms: Ancillary study group

SUMMARY:
Ischemic stroke is the first cause of acquired disability of the adult, the second cause of dementia and the third cause of death in the industrialized countries, what constitutes à major public health issue. Stroke is characterized by a cerebral parenchymal lesion due to an ischemic mechanism (85% of the cases) or hemorrhagic mechanism (15%). For a long time, the only approved treatment was the intravenous thrombolysis (rt-PA). Recently, thrombectomy has proven its superiority in this pathology.

Cohorts of patients with stroke are rare but can be very valuable by their clinical, laboratory and imaging well documented. They are the source of new hypotheses for research or interventions as well as the quality of care assessment tool.

The main objective of this project is to identify new markers: biological and imaging, treatment response and prognosis after ischemic stroke.

Secondary objectives of the HIBISCUS-STROKE II cohort are to establish a clinical database, completed by biological samples and by imaging data that can be used in the following areas:

Descriptive epidemiology of ischemic stroke and cerebral reperfusion, Pharmacoepidemiology and treatments observatory: safety, efficacy, indication of treatment in real life, costs Assessment of the long-term effect of the treatment on the occurrence of disability, stroke recurrence and death, Quality of life and personal, familial, professional and social consequences of stroke, Research of new diagnostic and prognostic biomarkers, Research projects.

Ancillary study :

Cardiac complications are the second leading cause of death after stroke. A close relationship between brain damage and heart complications, referred to as "neuro-cardiac syndrome" has been established. 20% of patients admitted for ischemic stroke present at least one major cardiac event, including acute coronary syndrome, heart failure and / or cardiac arrhythmia, within three months of the event, while 28% have a left ventricular ejection fraction less than 50%. However, the underlying pathological mechanisms remain unclear and the therapeutic targets unknown. To study these mechanisms, an ancillary study will be proposed to patient whom accepted to participate in the main project research.

The general objective of the ancillary study is to identify early markers of cardiac damage during ischemic stroke having benefited from mechanical recanalization by thrombectomy, and to improve the understanding of the pathophysiology at the origin of cardiac complications in the course of an ischemic stroke with the final objective of identifying new therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Ischemic Stroke confirmed by MRI
* Proximal arterial occlusion (M1 and/or M2)
* Eligible for thrombolysis and/or thrombectomy
* Informed consent signed by the patient or the next of kin
* Patient with a social security number

Ancillary Study Inclusion Criteria:

* Eligible for the Hibiscus stroke II cohort
* Ancillary study informed consent signed by the patient or the next of kin

Exclusion Criteria:

* Patients for whom it is known at the inclusion that follow-up at 3 months will not be possible at Pierre Wertheimer Hospital (Lyon, France)
* Patient with progressive or uncontrolled cancer.
* Deprivation of civil rights
* Pregnant woman or woman of childbearing age without proof of the absence of a current pregnancy
* For patients participating in the optional fecal library: factors leading to a potential change in microbiota (antibiotic therapy within 3 months, probiotic or rebiotic use within 3 months, ileo or gastrostomy, gastrointestinal resection surgery, bariatric or peptic ulcer surgery, Crohn's disease or chronic inflammatory bowel disease, helicobacter pylori gastric ulcer less than 1 year old, participation in a study that aims to modify the microbiota)

Ancillary Study Exclusion Criteria:

* Contraindication to MRI with gadolinium injection
* Contraindication to cardiac MRI (including inability to perform cardiac MRI)
* Patients with a glomerular filtration rate <30ml/min
* History of coronary artery disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-05-22 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Specific primary endpoint will be established for each sub-study based on data from the HIBISCUS-Stroke II cohort such as the Rankin score at 3 months. | At month 3
  This study will allow the realization of various research exploiting the data collected. Each study will defined its relevant primary endpoint. The primary endpoint will most often be the Modified Rankin Scale (mRS from 0 to 6 where 6 is the worst outcome) at 3 months or the vital status at 3 months.

SECONDARY OUTCOMES:
Population description (Age, sex, risk factors, comorbidity, etc.) | At day 5 (± 2 days) after une initial hospitalization
  Descriptive Epidemiology of the study population
Recanalization efficacy | During the procedure (endovascular treatment)
  The efficacy of revascularization will be evaluated by TICI Score (Thrombolysis In Cerebral Infarction). A grade of zero indicated a recanalization failure and a grade of 3 a complete recanalization.
Long-term hemorrhagic onset | Day 1 after une initial hospitalization
  ECASS (European Cooperative Acute Stroke Study) Scale evaluation which divides hemorrhagic transformation into four subtypes from hemorrhagic infarction type 1 (HI1) to parenchymal hematoma type 2 (PH2)
Degree of disability (mRS Score) | Up to 1 year
  Degree of disability: modified Rankin Score
Quality of life (EQ5D questionnaire) | At 3, 12 months
  The quality of life of the patient will be assessed through the EQ5D questionnaire
Research of potential new markers | At month 49
  Research of new markers such as inflammatory cytokines (IL-6, IL-8, IL-10).
Myocardial damage from the ischemic stroke | Day 6 (±2days)
  Assessment of the irreversible lesions due to myocardial ischemia evaluated on MRI at day 6
Levels of NTproBNP and troponin | Day 6 (±2days)
  NTproBNP and troponin level measurement
Research of potential new biomarkers | Day 6 (±2days)
  Research of potential new biomarkers such as marker of the hematoencephalic barrier damages (MMP9)
Evaluation of the fecal bacterial microbiological profile | At Day 1, at month 3
  Evaluation of the fecal microbiological profile by 16S sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pierre Wertheimer, GHE, Bron, France